CLINICAL TRIAL: NCT03573232
Title: Prevalence of Abnormal Postures in Parkinson's Disease: an Observational Multicenter Study
Brief Title: Prevalence of Abnormal Postures in Parkinson's Disease
Acronym: POSTUREinPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Michele Tinazzi, MD, PhD, M.D., Ph.D. Full Professor, Universita di Verona
Other Study IDs: Università di Verona
Record Dates: First submitted 2018-05-07; First posted 2018-06-29 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Pisa Syndrome; Camptocormia; Antecollis; Striatal deformities
MeSH Terms: conditions — Parkinson Disease; Camptocormia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postural abnormalities represent disabling and painful complications in patients with Parkinson's disease (PD). The stooped posture is a typical feature of PD but with advancing of disease more severe body abnormalities can affect people with PD. These deformities include Pisa syndrome, camptocormia, antecollis, scoliosis and striatal deformities related to hand (striatal hand) and/or toes (striatal toes).

DETAILED DESCRIPTION:
Postural abnormalities represent disabling and painful complications in patients with Parkinson's disease (PD). The first postural trunk deviation in PD was first described by James Parkinson himself and recognized as stooped simian appearance, with flexion of the hips and knees, and rounding of the shoulders. Although the stooped posture is a typical feature, more severe spinal misalignment (and deformities) can affect people with PD. These postural deformities include Pisa syndrome (PS), camptocormia (CP), antecollis (AC), scoliosis (S) and striatal deformities related to hand (striatal hand) and/or toes (striatal toes). The prevalence of these postural deformities is variable because several diagnostic criteria have been used to characterize each deformity. Recently, a consensus of diagnostic criteria has been reached in literature permitting us to better mapping the presence of these deformities in people with PD.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be considered enrolled after signing the consent form;
2. Diagnosis of Parkinson's disease;

Exclusion Criteria:

1. Concomitant neurologic diseases known to negatively affect posture;
2. A history of major spinal surgery or muscle and/or skeletal diseases;
3. Treatment with drugs potentially able to induce abnormal postures;
4. Clinical features consistent with a diagnosis of atypical parkinsonism;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the present multicenter study, consecutive outpatients with PD attending 7 movement disorders Italian tertiary centers (Verona, Ancona, Chieti, Pisa, Torino, Trieste, Roma) will be invited to participate. Participants will be considered enrolled after signing the consent form.
Sampling Method: Probability Sample
Enrollment: 794 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-10-07 (Estimated); Study Completion 2018-10-07 (Estimated)

PRIMARY OUTCOMES:
The prevalence of postural deformities | 1 day
  % of people with Parkinson's disease reporting Pisa syndrome, camptocormia, antecollis, scoliosis and striatal deformities related to hand (striatal hand) and toes (striatal toes).

SECONDARY OUTCOMES:
Data of birth | 1 day
  (day/month/year);
Sex | 1 day
  (male/female)
Body Mass Index | 1 day
  (score)
SPECIFIC EVALUATION FOR PATIENTS WITH PARKINSON'S DISEASE • Age at PD onset | 1 day
  (years)
Disease duration of PD | 1 day
  (years)
Modified Hoehn and Yahr (H&Y); | 1 day
  Total score of Modified Hoehn and Yahr staging scale. It evaluates the stage of Parkinson's disease. Range= 1 to 5. Higher values represent worse stages of disease.
Unified Parkinson's Disease Rating Scale (UPDRS); | 1 day
  The Unified Parkinson's Disease Rating Scale evaluates the motor and non-motor symptoms of Parkinson's disease. Range= 0 to 260. Higher values represent worse symptoms of disease.
PD phenotype | 1 day
  (rigid acinetic; tremor; mixed type)
Laterality of motor symptoms at PD onset | 1 day
  (right, left, bilateral);
Clinical asymmetry | 1 day
  (number of patients)
Quality of life by means of Parkinson's Disease Questionnaire-8; | 1 day
  Parkinson's Disease Questionnaire-8 evaluates quality of life in patients with Parkinson's disease. Range= 0 to 100. Higher values represent worse quality of life.
Latency between PD onset and start of antiparkinsonian therapy | 1 day
  (years)
Pharmacologic treatment at disease onset of PD | 1 day
  (levodopa; dopaminoagonists; L-Dopa + dopaminoagonist; other therapies)
Ongoing pharmacological therapy | 1 day
  (levodopa; dopaminoagonists; L-Dopa + dopaminoagonist; other therapies)
Levodopa equivalent daily dose | 1 day
  (mg)
Number of falls and direction | 1 day
  (number, anterior, posterior, right, left)
Comorbilities | 1 day
  (heart diseases, malignancies, diabetes, hypertension, mental disorders, obesity, metabolic disorders, cerebrovascular diseases, physical trauma)
Associated medical conditions | 1 day
  (osteoporosis, arthrosis, rheumatic diseases, otovestibular disorders)
Visual Analogue Scale (VAS) | 1 day
  Visual Analogue Scale evaluates pain intensity. Range= 0 to 10. Higher values represent higher pain intensity.
SPECIFIC EVALUATION FOR PATIENTS WITH ABNORMAL POSTURES Type of deformity | 1 day
  (Pisa syndrome, camptocormia, anterocollis, scoliosis, striatal deformities)
Degrees | 1 day
  (wall goniometer and pictures with software-based analysis)
Latency to develop one or more postural deformity after PD onset | 1 day
  (months)
Postural deformity duration | 1 day
  (years)
The pattern of postural deformity onset | 1 day
  (acute, subacute, chronic)
Postural deformity after drug modification | 1 day
  (yes/no)
Postural deformity awareness | 1 day
  (yes/no)
Head compensation | 1 day
  (in case of PS, CP, AC)
Neck head on trunk angle | 1 day
  (degrees)
Neck tilt angle | 1 day
  (degrees)
Head tilt angle | 1 day
  (degrees)
Gaze angle (in case of AC) | 1 day
  (degrees)
Ankle and hip flexion (in case of CP) | 1 day
  (degrees)
Sensory trick | 1 day
  (yes/no)
Postural deformity direction only for PS | 1 day
  (right/left)
The presence of metronome sign (in case of PS) | 1 day
  (yes, no)
Side of PD symptoms at onset and PS inclination | 1 day
  (ipsilateral, contralateral, bilateral)
Side of PD symptoms at onset and hands/feet deformities | 1 day
  (ipsilateral, contralateral, bilateral)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tinazzi, MD, PhD, Professor, Principal Investigator — Universita di Verona; Nicola Smania, MD, Professor, Study Chair — Universita di Verona; Marialuisa Gandolfi, MD, PhD, Study Chair — Universita di Verona; Christian Geroin, PhD, Study Chair — Universita di Verona
Locations (7):
- Italy (7):
  - Department of Experimental and Clinical Medicine - University "Politecnica delle Marche" Ancona -Italy. Neurorehabilitation Clinic - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona., Ancona
  - Department of Neuroscience, Imaging and Clinical Sciences, University G.d'Annunzio of Chieti-Pescara, Pescara
  - Neurology Unit, Department of Clinical and Experimental Medicine, University of Pisa, Pisa, Italy, Pisa
  - IRCCS San Raffaele CTC Centro Parkinson Via della Pisana 235, 00163 Roma, Roma
  - Dipartimento di Neuroscienze A.O. Città della Salute e della Scienza di Torino, Torino
  - Clinica Neurologica, Dipartimento di Scienze Neurologiche, Chirurgiche e della Salute, Azienda Ospedaliera Universitaria integrata, Universita' di Trieste, Trieste
  - Department of Neurosciences, Biomedicine and Movement Sciences, University of Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doherty KM, van de Warrenburg BP, Peralta MC, Silveira-Moriyama L, Azulay JP, Gershanik OS, Bloem BR. Postural deformities in Parkinson's disease. Lancet Neurol. 2011 Jun;10(6):538-49. doi: 10.1016/S1474-4422(11)70067-9. Epub 2011 Apr 22. PMID 21514890
- [Background] Tinazzi M, Geroin C, Gandolfi M, Smania N, Tamburin S, Morgante F, Fasano A. Pisa syndrome in Parkinson's disease: An integrated approach from pathophysiology to management. Mov Disord. 2016 Dec;31(12):1785-1795. doi: 10.1002/mds.26829. Epub 2016 Oct 25. PMID 27779784
- [Background] Srivanitchapoom P, Hallett M. Camptocormia in Parkinson's disease: definition, epidemiology, pathogenesis and treatment modalities. J Neurol Neurosurg Psychiatry. 2016 Jan;87(1):75-85. doi: 10.1136/jnnp-2014-310049. Epub 2015 Apr 20. PMID 25896683
- [Background] Pandey S, Garg H. Postural & striatal deformities in Parkinson;s disease: Are these rare? Indian J Med Res. 2016 Jan;143(1):11-7. doi: 10.4103/0971-5916.178577. PMID 26997007